CLINICAL TRIAL: NCT06201793
Title: Clinical Study to Evaluate the Possible Efficacy and Safety of Minocycline in Patients With Ulcerative Colitis Treated With Mesalamine
Brief Title: Minocyclin in Ulcerative Colitis as Added on Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mostafa Bahaa (Other)
Collaborators: Amira Fawzy Mohamed Mashaly, Clinical Pharmacy Demonstrator, Faculty of Pharmacy- Horus University (Unknown); Tanta University (Other); Mounir Hussein Bahgat Internal Medicine Department Mansoura University (Unknown)
Responsible Party: Sponsor-Investigator, Mostafa Bahaa, Teaching assisstant, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 236977
Record Dates: First submitted 2023-12-31; First posted 2024-01-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Mesalamine; Minocycline

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): control group (Mesalamine group, n =23) who will receive 1 g mesalamine three times daily for 6 months.
  Interventions: Drug: Mesalazine
- Minocycline group (Active Comparator): minocycline group, n = 23) will receive 1 g mesalamine three times daily plus 100 mg minocycline orally twice daily for 6 months.
  Interventions: Drug: Mesalazine; Drug: Minocycline

INTERVENTIONS:
Drug: Mesalazine — Mesalamine, also known as 5-aminosalicylic acid (5-ASA), is a medication used to treat ulcerative colitis. It is usually used to induce or maintain remission of mildly to moderately active ulcerative colitis
Drug: Minocycline — Minocycline is a tetracycline antibiotic medication used to treat a number of bacterial infections such as pneumonia. It is generally less preferred than the tetracycline doxycycline. Minocycline is also used for the treatment of acne and rheumatoid arthritis.
  Arms: Minocycline group

SUMMARY:
Ulcerative colitis (UC) is considered a subcategory of inflammatory bowel disease and the exact cause of ulcerative colitis remains undetermined. the condition appears to be related dysregulated immune response and consequent activation of inflammatory cascades, which are often affected by genetic susceptibility and environmental factors, and 20% to 40% of patients with UC also exhibit extraintestinal manifestations involving the joints, skin, eyes, or hepatobiliary tract

DETAILED DESCRIPTION:
Most conventional UC therapies rely primarily on downregulating aberrant immune responses and inflammatory cascades. Mesalamine and corticosteroids are the mainstays in management of UC. However, 20% to 32% of UC patients do not respond to steroid.4 Some antibiotics offer protection against experimental and clinical colitis.

Mesalazine (also known as mesalamine or 5- amino salicylic acid, 5-ASA) has a well-established role in UC management. It is the first line therapy for mild to moderate UC and it is considered the cornerstone in the management of UC. The mechanism of action of mesalazine is diverse. It acts locally on colonic mucosa and reduce inflammation by several anti-inflammatory processes. It has a potent antioxidant and free-radical scavenger properties.

Nitrosative stress caused by inducible nitric oxide synthase (iNOS)-derived nitric oxide (NO) production and matrix metalloproteinases (MMPs) have been shown to play an important role in the pathogenesis of UC. As in human UC, expression of MMPs and iNOS are also implicated in the pathogenesis of experimental colitis, Therefore, it is important to develop and evaluate agents that have low-severity adverse effects that can treat UC by blocking inflammatory responses involved in nitrosative stress and/or MMP activation.

Minocycline, a semisynthetic tetracycline, is a safe, widely used and inexpensive antibiotic with a broad spectrum.

Several recent studies have demonstrated that, in addition to its antimicrobial effects, minocycline exerts anti-inflammatory, antiangiogenic, and antiapoptotic effects. These biological effects of minocycline have been shown to have a therapeutic or preventive effect in neurodegenerative disease, neural ischemic damage, ischemic renal injury, rheumatoid arthritis, acne vulgaris, pyoderma gangrenosum, and periodontitis. The mechanisms by which minocycline alleviates these illnesses involve suppressing expression and/or activity of iNOS, MMPs, TNF-α and caspases, and blocking cytochrome-c release. Several animal models of intestinal inflammation have been established, although some only partially resemble human UC.

Also, minocycline improved the colonic oxidative status and decreased the expression of different chemotactic mediators like expressions of the chemokine's monocyte chemotactic protein-1 (MCP-1) and cytokine-induced neutrophil chemoattractant-1 (CINC-1) as well as of the intercellular adhesion molecule-1 (ICAM-1) in the inflamed tissue. However, the in vitro experiments performed revealed that minocycline reduced the release of the chemokine IL-8 by the intestinal epithelial cells Caco-2.

The immunological activity of minocycline was reinforced by its remarkable effect in restoring a balanced intestinal microbiota. the preclinical study shows that the counts of lactobacilli and bifidobacteria, which were downregulated in colitic rats from control group when compared with healthy rats, only appeared increased after treatment with minocycline.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years old Both male and female will be included Mild and moderate UC patients diagnosed and confirmed by endoscope Patient treated with 5-aminosalislic acid (mesalamine)

Exclusion Criteria:

Patients with severe UC Pregnancy and lactating females Significant liver and kidney function abnormalities Diabetic patients Patients with Colorectal cancer patients Patients taking rectal or systemic steroids Patients on immunosuppressants or biological therapies Patients taking antacids, anticoagulants, bactericidal antibiotics, oral contraceptives, and isotretinoin.

Addiction to alcohol and / or drugs Known allergy to the studied medications History of complete or partial colectomy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Assessment of disease activity using Partial Mayo Scoring Index | 6 months
  Partial Mayo Scoring Index (PMSI) assessment for Ulcerative Colitis Activity. It depends on three items; stool frequency, rectal bleeding (blood in stool) and Physician's Global Assessment. Each item has a score from 0 to 3 and total PMSI is the sum of scores for the three items.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Derived] Mashaly AF, Hegazy SK, Bahgat MM. Repurposing minocycline as an added-on treatment for ulcerative colitis patients on mesalamine: a randomized clinical pilot study. Naunyn Schmiedebergs Arch Pharmacol. 2025 Oct 23. doi: 10.1007/s00210-025-04662-2. Online ahead of print. PMID 41128897